CLINICAL TRIAL: NCT02193217
Title: A Phase 1 Study to Explore the Cardiac Pharmacodynamics of MT-1303
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-1303-E12
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

ARMS (4):
- MT-1303-Low (Experimental): MT-1303-Low dose
  Interventions: Drug: MT-1303-Low
- MT-1303-High (Experimental): MT-1303-High dose
  Interventions: Drug: MT-1303-High
- Fingolimod (Active Comparator): Fingolimod
  Interventions: Drug: Fingolimod
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-1303-Low
  Arms: MT-1303-Low
Drug: MT-1303-High
  Arms: MT-1303-High
Drug: Fingolimod
  Arms: Fingolimod
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the cardiac pharmacodynamics, safety and tolerability of MT-1303 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease.
* Male and female subjects of non-childbearing potential aged 18 to 55 years.
* Normal or non-clinically significant 12-lead ECG.
* Holter recording with no clinically significant abnormalities.
* Systolic blood pressure: 90 to 140 mmHg, diastolic blood pressure: 50 to 90 mmHg

Exclusion Criteria:

* A History of severe adverse reaction or allergy to any medical product.
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastrointestinal, renal, cardiovascular disease, eye disorder or history of psychiatric/psychotic disorder.
* A history of tuberculosis.
* Have a positive HBsAg, HBcAb, HCVAb or HIV-1 and HIV-2 test.
* Previously having received MT-1303, fingolimod, or any other sphingosine-1-phosphate receptor modulators.
* Clinical relevant abnormal medical history, or physical findings or laboratory values.
* Clinically significant 12-lead ECG abnormalities.
* Clinical relevant abnormal findings in echocardiograph.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mean hourly heart rate | up to day 42

SECONDARY OUTCOMES:
Plasma concentration of MT-1303 and its metabolite | up to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sowood, M.D, Study Director — Mitsubishi Tanabe Pharma Europe Ltd.
Locations (1):
- Investigational site, Leeds, United Kingdom